CLINICAL TRIAL: NCT05067491
Title: Bringing Exposure Therapy for Animal Phobias to Real-Life Context With Augmented Reality-Dogs
Brief Title: Bringing Exposure Therapy to Real-Life Context With Augmented Reality-Dogs (ARET)-Dogs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Arash Javanbakht, Director of Stress, Trauma, and Anxiety Research Clinic, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1711000968-Dog Phobia
Record Dates: First submitted 2021-09-21; First posted 2021-10-05 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Specific Phobia, Animal
Keywords: Exposure therapy; Technology; Telemedicine; Cynophobia
MeSH Terms: conditions — Phobia, Specific; Zoophobia

STUDY DESIGN:
Intervention Model Description: 15 Intervention vs 15 non-intervention control group for cynophobia (fear of dogs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The experimental group will go through an exposure therapy session using an augmented reality headset device. The participant will work with the therapist, who will control the augmented reality paradigm and cater the exposure to the needs of the participant. The duration of the exposure will be as long as is needed to reduce anxiety regarding the feared object until self-reported subjective distress is low and stable.
  Interventions: Behavioral: Augmented reality exposure therapy
- Non-intervention (No Intervention): The control group will not go through an exposure therapy session using an augmented reality headset device. This will be a no-intervention control group that can have some form of exposure therapy following the conclusion of the treatment/research period.

INTERVENTIONS:
Behavioral: Augmented reality exposure therapy — Virtual objects will be placed in the patient's visual field, superimposed on their real environment for exposure therapy.
  Other Names: Exposure therapy via utilization of augmented reality
  Arms: Intervention

SUMMARY:
In this patented project, U.S. Patent No. 10,839,707, the investigators will develop an augmented reality exposure therapy method for cynophobia, also known as dog phobia, to test in the clinic. The platform will include a software that allows the clinician (psychiatrist/therapist) to position virtual objects in the real environment of the patient with the above mentioned phobia while the patient is wearing the augmented reality (AR) device. Then the clinician will lead the patient through steps of exposure therapy to the feared object. The investigators will then measure the impact of treatment and compare to before treatment measures of fear of the phobic object.

Exposure therapy is the most evidence-based treatment for specific phobias, social phobia, obsessive-compulsive disorder (OCD), and posttraumatic stress disorder (PTSD). The core principle is patient's exposure to the feared objects/situations guided by a clinician. For example, in cynophobia, patient is exposed to pictures of dogs printed or on a computer screen - or if available, view of a real dog in the office. Gradually, patient tolerates viewing/approaching the dog from a closer distance, and fear response extinguishes. The clinician has a crucial role in signaling safety to the patient, as well as providing support and coaching. This treatment is limited by multiple factors: 1) limited access to feared objects/situations in the clinic, 2) even when feared objects are available, they are not diverse (e.g. different types, sizes, and colors of dogs), which limits generalization of safety learning, 3) when available, clinician has very limited control over behaviors of the feared object, 4) safety learning is limited to the clinic office context, and contextualization of safety learning to real life experiences is left to the patient to do alone, which often does not happen. This is specifically important in conditions such as PTSD, where there is cumulative evidence for impaired contextualization as a key neurobiological underpinning. 5) Lack of geographical access to experts in exposure therapy, especially for PTSD, in rural areas.

DETAILED DESCRIPTION:
Anxiety and stress-related disorders are very common. One in three people experience some form of anxiety disorder including phobias, PTSD, and OCD. These disorders chronically limit one's ability to function and enjoy life. In addition to the common prevalence, wars in Iraq and Afghanistan have left about 13% of the returning veterans with combat PTSD, and even more with partial symptoms. Lifetime prevalence of PTSD is as high as 10% in women. Economic burden of anxiety disorders is between 42 to 52 billion dollars, one third of the country's total mental health bill. Near 30% of this money is spent in treatment costs. Burden of lost workdays only for PTSD is $3 billion.

Exposure therapy is the most effective treatment for cue-related anxiety disorders such as specific phobias, social phobia, OCD, and PTSD. The core principle is exposure to the feared objects/situations guided by a clinician. For example, in cynophobia (fear of dogs) patient is exposed to picture of a dog on a computer, or from distance in the office, and gradually, with help of the clinician, they tolerate view of the dog from a closer distance. Clinician has a crucial role as the social safety cue in this process.

Although exposure therapy is very effective in treatment of phobias, OCD, and PTSD, there are limitations. Access and adherence to, and efficacy of exposure therapy are limited to 50% by multiple factors: First, there is a national shortage of psychiatrists and psychotherapists; patients often have to be on waiting list for weeks to months, and in many geographical locations such services are extremely scarce or do not exist. More than 50% of clinicians are not trained in exposure therapy, and there is usually geographical barriers for access to skilled therapists. In general, more than half of the US counties are unable to recruit mental health providers. Very frequently patients only receive medication or supportive therapy for several years before they can see a specialist trained in exposure therapy. Certain conditions like social phobia or PTSD make it increasingly difficult to leave the house and go to the clinic. Second, the feared objects are not always available in office for exposure and exposure most of the times is limited to pictures, movie clips, imagination, narrative, or memories. Imaginary exposure commonly lacks the level of arousal that is required for development of new safety learning. Third, patients have to practice real-life exposure on their own. In vivo treatment is commonly limited: often patients do not create situations that elicit the optimal safety learning, do not know how to create exposure situations, or simply do not follow through because of high anxiety in the absence of someone to coach them. This gap between exposure in the office, and real-life exposure remains a significant roadblock in successful exposure therapy. Fourth, clinicians are usually unable to provide treatment across multiple physical, temporal and social contexts that can promote contextualization of safety learning. Exposure mostly happens in the physical, emotional, social, and temporal context of the office visits. A fifth limitation is that current exposure therapy methods, do not address overgeneralization of the fear response.

Augmented Reality Augmented reality (AR) is the next wave of interactive human-computer technology that provides an opportunity of mixing virtually created objects with reality. Instead of creating a completely synthetic environment, AR adds virtually created objects to the real non-synthetic context. These elements become part of the real context, or cover some of its components. AR technology ultimately becomes less expensive than virtual reality (VR) technology because it does not require modeling the whole environment.

The investigators developed a proof of concept prototype. The prototype includes a scenario for treatment of fear of spiders (arachnophobia). The software platform connects the patient to a clinician who is located in the same or a different physical space, the patient wears the AR device, the clinician is able to see the patient's field of view, and positions a virtual spider on a surface in the patient's environment, clinician determines direction/velocity of motions of the virtual spider, clinician leads patient through the process of exposure therapy process until patient is desensitized to the view of the spider. Exposure can then advance to higher number of spiders, or larger ones. After successful use of the spider prototype, the investigators have developed a program for use with cynophobic patients.

Subject Recruitment: Subject recruitment will happen at the Wayne State University (WSU) Department of Psychiatry and Behavioral Neurosciences (DPBN) psychiatry clinic, through flyers spread on the campus, and advertisement on Wayne State's student website. The investigators aim to pre-screen a minimum of 50 individuals. The actual number of participants to be enrolled is 40, and the investigators have a minimum pre-screening of 50 anticipating that some may not qualify.

Treatment will take place at the Stress, Trauma, and Anxiety Research Clinic at the WSU department of psychiatry in Detroit. Participants will do 1-4 sessions of augmented reality exposure therapy (ARET), each lasting up to 90 minutes. The first session will include a short refresher on principles of exposure therapy, and training the use of the AR equipment. Treatment is concluded when the patient is stably showing Subjective Units of Distress (SUDs) < 4 to the maximum level of AR exposure to virtual dogs.

At any time the level of distress due to exposure is determined too high, both patient and the provider can abort the exposure. This will be done similarly to any other conventional exposure therapy method.

ELIGIBILITY:
Inclusion Criteria:

Primary diagnosis of dog phobia, according to Diagnostic and Statistical Manual-5 (DSM-5) criteria

Willing and able to consent for involvement in the study

Exclusion Criteria:

People who refuse or are unable to consent to participate in the study

Current or previous diagnosis of psychotic disorder, schizophrenia, bipolar disorder, PTSD, mental retardation, active abuse of substances or meet criteria for substance use disorder in the past six months

Unstable behavior that, in the opinion of the investigator, would place the participant at increased risk or preclude the participant's full compliance with or completion of the study, e.g., significant Axis II disorder or suicidal behavior

Visual or auditory disabilities limiting ability to use the AR goggles

Current use of antidepressant medications, mood stabilizers, or benzodiazepines

History of seizures or a condition that would increase likelihood for seizures

Serious medical or neurological illness

Wards of the court

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Behavioral Approach Test--Ability to confront phobia | Change in score on Behavioral Approach Test from baseline to post treatment (immediately following the last exposure therapy session and at one-month follow-up)
  A measure of the closest distance the patient can have to the feared object. Scored from 0-12 based on distance away from feared object and interaction with feared object. The score is given based on participant interaction, therefore one value is chosen. Higher values closer to 12 show greater comfortability and ability to interact with the feared object.

SECONDARY OUTCOMES:
Cynophobia (fear of dogs) as measured by the Dog Phobia Questionnaire (DPQ) | Change in score on Dog Phobia Questionnaire from baseline to post treatment (immediately following the last exposure therapy session and at one-month follow-up)
  The DPQ is a 27-item, self-report questionnaire designed to measure symptoms of dog phobia. Respondents are asked to "indicate the degree to which you agree or disagree with each statement as it applies to you in the past month" using a 7-point Likert-type scale, with anchors of 1 ("strongly agree"), 4("neutral"), and 7 ("strongly agree"). Four items are reverse scored (e.g., "I would not feel nervous if I saw a dog"). The scale yields a minimum score of 27 and a maximum score of 189.

OTHER OUTCOMES:
Autonomic Arousal | Change in score from baseline to post treatment (immediately following the last exposure therapy session and at one-month follow-up)
  Galvanic skin response will be used to assess hyperarousal throughout the sessions. Galvanic skin response will be measured as the magnitude of the change from baseline to presentation of feared stimulus. Higher Skin Conductance Response (SCR) is associated with greater autonomic arousal/fear of the object.
Credibility and expectancy of treatment efficacy as measured by the Credibility/Expectancy Questionnaire | Change in score from baseline to post treatment (immediately following the last exposure therapy session and at one-month follow-up)
  The Credibility/Expectancy questionnaire is 6 items scored on a scale from 1-9, for a low score of 6 and a high score of 54. Total score is calculated by adding all items together. Higher scores are indicative of greater expectancy in treatment credibility and efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Arash Javanbakht, MD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University Department of Psychiatry and Behavioral Neurosciences, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Botella C, Perez-Ara MA, Breton-Lopez J, Quero S, Garcia-Palacios A, Banos RM. In Vivo versus Augmented Reality Exposure in the Treatment of Small Animal Phobia: A Randomized Controlled Trial. PLoS One. 2016 Feb 17;11(2):e0148237. doi: 10.1371/journal.pone.0148237. eCollection 2016. PMID 26886423
- [Background] Wrzesien M, Burkhardt JM, Alcaniz Raya M, Botella C, Breton Lopez JM. Analysis of distributed-collaborative activity during augmented reality exposure therapy for cockroach phobia. Stud Health Technol Inform. 2010;154:134-9. PMID 20543285
- [Background] Foa EB, McLean CP. The Efficacy of Exposure Therapy for Anxiety-Related Disorders and Its Underlying Mechanisms: The Case of OCD and PTSD. Annu Rev Clin Psychol. 2016;12:1-28. doi: 10.1146/annurev-clinpsy-021815-093533. Epub 2015 Nov 11. PMID 26565122
- [Background] Tarrier N, Pilgrim H, Sommerfield C, Faragher B, Reynolds M, Graham E, Barrowclough C. A randomized trial of cognitive therapy and imaginal exposure in the treatment of chronic posttraumatic stress disorder. J Consult Clin Psychol. 1999 Feb;67(1):13-8. doi: 10.1037//0022-006x.67.1.13. PMID 10028204
- [Background] Tsai CF, Yeh SC, Huang Y, Wu Z, Cui J, Zheng L. The Effect of Augmented Reality and Virtual Reality on Inducing Anxiety for Exposure Therapy: A Comparison Using Heart Rate Variability. J Healthc Eng. 2018 Nov 25;2018:6357351. doi: 10.1155/2018/6357351. eCollection 2018. PMID 30595830
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Vorstenbosch V, Antony MM, Koerner N, Boivin MK. Assessing dog fear: evaluating the psychometric properties of the Dog Phobia Questionnaire. J Behav Ther Exp Psychiatry. 2012 Jun;43(2):780-6. doi: 10.1016/j.jbtep.2011.10.006. Epub 2011 Oct 28. PMID 22104660